CLINICAL TRIAL: NCT02589275
Title: A 3-Month, Multicenter, Open-Label Extension to Evaluate Safety and Efficacy of TNX-102 SL Tablets Taken Daily at Bedtime in Patients With Fibromyalgia
Brief Title: A 3-Month Open-Label Safety and Efficacy Study of TNX-102 SL Tablets in Fibromyalgia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-F303
Record Dates: First submitted 2015-10-19; First posted 2015-10-28 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Primary Fibromyalgia
Keywords: TNX-102 SL; bedtime; sublingual; 3-month; long term safety; long term efficacy; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TNX-102 SL Tablet 2.8 mg (Experimental): 1x TNX-102 SL 2.8 mg sublingual tablet taken daily at bedtime for 3 months
  Interventions: Drug: TNX-102 SL Tablet 2.8 mg

INTERVENTIONS:
Drug: TNX-102 SL Tablet 2.8 mg — TNX-102 SL 2.8 mg tablet taken daily at bedtime
  Other Names: cyclobenzaprine

SUMMARY:
This is a Phase 3, open-label, extension trial designed to evaluate the long term safety and efficacy over 3 months of TNX-102 SL tablets taken daily at bedtime for the treatment of Fibromyalgia (FM). Patients recruits into this trial are those who have successfully completed the double-blind studies; TNX-CY-F301 and TNX-CY-F302.

Patients will not be made aware of the therapy they received during the double-blind study.

DETAILED DESCRIPTION:
The study consist of 4 study visits, including Screening/Baseline Visit 1 (Day 1, which is anticipated to be the same date as Visit 6 in F301 or F302) and visits after 1, 2 and 3 months of treatment (Visits 2-4).

Primary:

The primary objective of the study is to evaluate the safety of TNX-102 SL tablets taken daily at bedtime over an additional 3 months in patients with FM who have completed the double-blinded lead-in study

Secondary:

The secondary objective is to evaluate the efficacy of TNX-102 SL tablets taken daily at bedtime to control symptoms of FM

ELIGIBILITY:
Inclusion Criteria:

* The patient met all prior inclusion and exclusion requirements for study F301 or F302 originally, and has had no intervening medical conditions, increased suicidal ideation, or requirements for concomitant medications that preclude exposure to TNX-102 SL or enrollment in the extension study.
* The patient completed expected dosing in F301 or F302 defined as taking study medication up to Week 12, with at least 70% compliance with medication usage (based on overall drug accountability reconciliation at the end of the F301 or F302 lead-in study) and no major protocol deviations.
* The patient has provided written informed consent to participate in this extension protocol.

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Sacramento, California
  - San Diego, California
  - Brandon, Florida
  - DeLand, Florida
  - Lakeland, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Smyrna, Georgia
  - Evansville, Indiana
  - North Dartmouth, Massachusetts
  - Ann Arbor, Michigan
  - Jackson, Mississippi
  - Williamsville, New York
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Warwick, Rhode Island
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Dallas, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- TNX-TNX: This group received 1x 2.8 mg TNX-102 SL sublingual tablet daily in the lead in study TNX-CY-F301, then continued to receive 1x 2.8 mg TNX-102 SL sublingual tablet in this open-label extension study.
- PBO-TNX: This group received 1x Placebo sublingual tablet daily in the lead in study TNX-CY-F301, then received 1x 2.8 mg TNX-102 SL sublingual tablet in this open-label extension study.
Period: Overall Study
Arm/Group | TNX-TNX | PBO-TNX
Started | 177 | 198
Completed | 143 | 142
Not Completed | 34 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNX-TNX | PBO-TNX | Total
Number analyzed (Participants) | 177 | 198 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (11.35) | 48.0 (10.77) | 48.1 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 191 | 360
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 19 | 25
  White | 166 | 172 | 338
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 177 | 198 | 375

OUTCOME MEASURES:

1. Primary Outcome: Newly Emergent Adverse Events
Description: The number of patients with at least one adverse event which began after the first dose of TNX-102 SL in this open-label extension study.
Time Frame: Up to 3 months from first dose
Population: Data is reported for all patients with AE data collected at the time when this study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | TNX-TNX | PBO-TNX
Number analyzed (Participants) | 170 | 186
Participants | 77 | 132

ADVERSE EVENTS:
Time Frame: Up to 3 months from first dose.
Description: All-cause mortality is reported for all patients. For AEs and SAEs, data is reported for all patients with AE data collected at the time when this study was terminated.
Arm/Group | TNX-TNX | PBO-TNX
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/198
Serious Adverse Events (participants affected / at risk) | 2/170 | 0/186
Other Adverse Events (participants affected / at risk) | 69/170 | 86/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-TNX (N=170) | PBO-TNX (N=186)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TNX-TNX (N=170) | PBO-TNX (N=186)
Hypoaesthesia Oral (Gastrointestinal disorders) | 60 | 73
Parasthesia Oral (Gastrointestinal disorders) | 9 | 11
Tongue Discomfort (Gastrointestinal disorders) | 5 | 15
Product Taste Abnormal (Product Issues) | 9 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all study investigators.